CLINICAL TRIAL: NCT05637476
Title: Effect of Functional Strength Training of Hip Abductors in Runners With Medial Tibial Stress :(Randomised Clinical Trail)
Brief Title: Effect of Functional Strength Training of Hip Abductors in Runners With Medial Tibial Stress Syndrome
Acronym: MTSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shreen Lashien, Senior musculoskeletal physiotherapist ,faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Medial tibial stress syndrome
Record Dates: First submitted 2022-11-13; First posted 2022-12-05 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Medial Tibial Stress Syndrome
Keywords: Recreational runners; Frontal plane projection angle; Pelvic drop height; Kinovea software
MeSH Terms: conditions — Medial Tibial Stress Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active control group) (Active Comparator): Group A (number=20): which is the control group with medial tibial stress syndrome, they will receive a selected physical therapy exercise program.
  Interventions: Other: A selected physical therapy exercise program
- Group B (Experimental group) (Experimental): Group B (number=20): which is the experimental group with Medial tibial stress syndrome, they will receive the same physical therapy exercise program as group A in addition to, functional strength training of hip abductors.
  Interventions: Other: Functional strength training of hip abductors; Other: A selected physical therapy exercise program

INTERVENTIONS:
Other: Functional strength training of hip abductors — Every participant will perform three sets of fifteen repetitions, fifteen seconds rest in between, three times per week for the following exercises:
  1. Pelvic drop.
  2. Single leg -bridge.
  3. Side-lying hip abduction with hip internal rotation.
  4. Lateral step-up.
  5. Standing hip abduction on stance or swing leg with extra resistance .
  Arms: Group B (Experimental group)
Other: A selected physical therapy exercise program — Every participant will perform three sets of fifteen repetitions, fifteen seconds rest in between, three times per week for the following exercises:
  1. Strength dorsiflexors of the ankle-using rubber band.
  2. Eccentric calf exercise (calf raise) .
  3. Balance and proprioceptive exercise using wobble boards.
  4. Stretch planter flexors (three sets of thirty repetitions, thirty seconds rest in between, three times per week)
  Other Names: Common established treatment exercises

SUMMARY:
This study will be the first project to investigate the effect of functional strength training of hip abductors on pain, function, hip, and knee kinematics including contra-lateral pelvic drop angle (hip frontal plane projection angle) and dynamic knee valgus (knee frontal plane projection angle) in runners with medial tibial stress syndrome patients.

DETAILED DESCRIPTION:
Forty participants with medial tibial stress syndrome will be recruited from orthopedic out clinic of the faculty of Physical therapy, Cairo, University, and Gezira Youth Center. They will be asked to sign the informed consent form .

The selected participants will be randomly assigned to two groups using a simple randomization method to allocate participants to the groups through the available online website www.randomization.com considering the control group as active control group. A flow diagram according to the Consolidated Standards of Reporting Trials (CONSORT) statement will be presented to illustrate the progression of this clinical trial .

Sample size calculation was performed using G*POWER statistical software (version 3.1.9.2; Franz Faul, Universitat Kiel, Germany) based on data of knee valgus angle derived from Pourahmad et al., (2021) who investigated the effect of strengthening the abductor and external rotator on lower limb kinematics in volleyball players with patellofemoral complications. The sample size required for this study was approximately 15 subjects in each group. Calculation is made with α=0.05, power = 80% and effect size = 1.1. The sample size increased to 18 subjects per group for possible dropout of 20%.

For statistical analysis:

* Unpaired t-test will be conducted for comparison of the subject characteristics between groups.
* Chi- squared test will be conducted for comparison of sex distribution between groups.
* Mixed MANOVA will be conducted to investigate the effect of treatment on pain, function, contralateral pelvic drop angle and dynamic knee valgus.
* Post-hoc tests using the Bonferroni test were carried out for subsequent multiple comparison.
* Statistical measures will be performed through the statistical package for social studies (SPSS) version 25 for windows.
* The level of significance for all statistical tests will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Athletes (runners) with a referred diagnosis of MTSS for at least 1 month
* Participants with bilateral affection, the most affected limb will be included in measurements.
* Body mass index range between (18.5-25 kg /m2 )

Exclusion Criteria:

* History of previous lower extremity surgery
* Neurological problems that will affect lower extremity function
* Recent or old fractures at lower limbs
* Cognitive impairment
* Medications (anti-inflammatory/muscle relaxant)
* Tumours

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The Frontal Plane Projection Angle | Change from baseline frontal plane projection angle at 8 weeks.
  It is a measure of the degree of dynamic knee valgus during functional tasks. FPPA is an angle that consists of two lines. One line between the thigh and hip markers and the other line between the ankle and knee markers .So that,from a frontal view, when the knee marker is medial to a line from the ankle marker to the thigh marker,the FPPA is negative (knee valgus).While,The FPPA is positive if the knee marker is lateral to a line drawn from ankle marker to the thigh marker (knee varus).
The contra-lateral pelvic drop angle | Change from baseline contra-lateral pelvic drop angle at 8 weeks.
  It is determined as the angle subtended by one line connecting the anterior superior iliac spine with the stance and swing limb and a second line drawn perpendicular to the stance limb anterior superior iliac spine then, the measurement will be subtracted from 90 degrees.

SECONDARY OUTCOMES:
Pain severity | 8 weeks
  Through using the visual analogue scale to detect the change from the baseline pain severity at eight weeks exercises treatment program. The participant will be asked to assess the worst pain level experience at last three days. The pain visual analogue scale is a uni-dimensional measure of pain severity,a straight horizontal line of fixed length,usually 10 cm.Using a ruler, the score is determined by measuring the distance (mm)on the 10-cm line between the no pain anchor and the patient's mark,providing a range of scores from 0-100. A higher score indicates greater pain intensity,while a lower score indicates lesser pain
Lower extremity function | 8 weeks
  Through using the lower extremity functional scale to detect the change from the baseline lower extremity function at eight weeks exercises treatment program.It is a self-report questionnaire.Twenty questions that assesses a person's capacity doing twenty different everyday activities.Patients select an answer from the following scale for each activity listed:
  1. Extreme difficulty.
  2. Quite a bit of difficulty.
  3. Moderate difficulty.
  4. A little bit of difficulty.
  5. No difficulty.
  Scoring guidelines to determine the final score,the scale's columns are added together, thus, the maximum possible score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function.While 9 scale points are the smallest difference that may be seen and the smallest variation that is clinically significant.Percentage of maximum function=(lower extermity function scale score)/80*100.

CONTACTS AND LOCATIONS:
Overall Officials: Ebtessam F Gomaa, Doctorate, Study Chair — Cairo University
Locations (1):
- Orthopedic out clinic of the faculty of Physical therapy, Cairo, University,and Gezira Youth Center., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson RL, Nee RJ. Analysis of hip strength in females seeking physical therapy treatment for unilateral patellofemoral pain syndrome. J Orthop Sports Phys Ther. 2007 May;37(5):232-8. doi: 10.2519/jospt.2007.2439. PMID 17549951
- [Result] Irawan DS, Huoth C, Sinsurin K, Kiratisin P, Vachalathiti R, Richards J. Concurrent Validity and Reliability of Two-dimensional Frontal Plane Knee Measurements during Multi-directional Cutting Maneuvers. Int J Sports Phys Ther. 2022 Feb 2;17(2):148-155. doi: 10.26603/001c.31651. eCollection 2022. PMID 35136683
- [Result] Almeida GP, Silva AP, Franca FJ, Magalhaes MO, Burke TN, Marques AP. Q-angle in patellofemoral pain: relationship with dynamic knee valgus, hip abductor torque, pain and function. Rev Bras Ortop. 2016 Feb 9;51(2):181-6. doi: 10.1016/j.rboe.2016.01.010. eCollection 2016 Mar-Apr. PMID 27069887
- [Result] Cashman GE. The effect of weak hip abductors or external rotators on knee valgus kinematics in healthy subjects: a systematic review. J Sport Rehabil. 2012 Aug;21(3):273-84. doi: 10.1123/jsr.21.3.273. PMID 22894982
- [Result] Chuter VH, Janse de Jonge XA. Proximal and distal contributions to lower extremity injury: a review of the literature. Gait Posture. 2012 May;36(1):7-15. doi: 10.1016/j.gaitpost.2012.02.001. Epub 2012 Mar 21. PMID 22440758
- [Result] Cichanowski HR, Schmitt JS, Johnson RJ, Niemuth PE. Hip strength in collegiate female athletes with patellofemoral pain. Med Sci Sports Exerc. 2007 Aug;39(8):1227-32. doi: 10.1249/mss.0b013e3180601109. PMID 17762354
- [Result] Craig DI. Medial tibial stress syndrome: evidence-based prevention. J Athl Train. 2008 May-Jun;43(3):316-8. doi: 10.4085/1062-6050-43.3.316. PMID 18523568
- [Result] Dierks TA, Manal KT, Hamill J, Davis IS. Proximal and distal influences on hip and knee kinematics in runners with patellofemoral pain during a prolonged run. J Orthop Sports Phys Ther. 2008 Aug;38(8):448-56. doi: 10.2519/jospt.2008.2490. Epub 2008 Aug 1. PMID 18678957
- [Result] Ferber R, Davis IM, Williams DS 3rd. Gender differences in lower extremity mechanics during running. Clin Biomech (Bristol). 2003 May;18(4):350-7. doi: 10.1016/s0268-0033(03)00025-1. PMID 12689785
- [Result] Franklyn M, Oakes B. Aetiology and mechanisms of injury in medial tibial stress syndrome: Current and future developments. World J Orthop. 2015 Sep 18;6(8):577-89. doi: 10.5312/wjo.v6.i8.577. eCollection 2015 Sep 18. PMID 26396934
- [Result] Galbraith RM, Lavallee ME. Medial tibial stress syndrome: conservative treatment options. Curr Rev Musculoskelet Med. 2009 Oct 7;2(3):127-33. doi: 10.1007/s12178-009-9055-6. PMID 19809896
- [Result] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Result] Hreljac A, Marshall RN, Hume PA. Evaluation of lower extremity overuse injury potential in runners. Med Sci Sports Exerc. 2000 Sep;32(9):1635-41. doi: 10.1097/00005768-200009000-00018. PMID 10994917
- [Result] Ireland ML, Willson JD, Ballantyne BT, Davis IM. Hip strength in females with and without patellofemoral pain. J Orthop Sports Phys Ther. 2003 Nov;33(11):671-6. doi: 10.2519/jospt.2003.33.11.671. PMID 14669962
- [Result] Leetun DT, Ireland ML, Willson JD, Ballantyne BT, Davis IM. Core stability measures as risk factors for lower extremity injury in athletes. Med Sci Sports Exerc. 2004 Jun;36(6):926-34. doi: 10.1249/01.mss.0000128145.75199.c3. PMID 15179160
- [Result] Mehta SP, Fulton A, Quach C, Thistle M, Toledo C, Evans NA. Measurement Properties of the Lower Extremity Functional Scale: A Systematic Review. J Orthop Sports Phys Ther. 2016 Mar;46(3):200-16. doi: 10.2519/jospt.2016.6165. Epub 2016 Jan 26. PMID 26813750
- [Result] Menendez C, Batalla L, Prieto A, Rodriguez MA, Crespo I, Olmedillas H. Medial Tibial Stress Syndrome in Novice and Recreational Runners: A Systematic Review. Int J Environ Res Public Health. 2020 Oct 13;17(20):7457. doi: 10.3390/ijerph17207457. PMID 33066291
- [Result] Fredericson M, Bergman AG, Hoffman KL, Dillingham MS. Tibial stress reaction in runners. Correlation of clinical symptoms and scintigraphy with a new magnetic resonance imaging grading system. Am J Sports Med. 1995 Jul-Aug;23(4):472-81. doi: 10.1177/036354659502300418. PMID 7573660
- [Result] Willson JD, Davis IS. Utility of the frontal plane projection angle in females with patellofemoral pain. J Orthop Sports Phys Ther. 2008 Oct;38(10):606-15. doi: 10.2519/jospt.2008.2706. PMID 18827327
- [Result] Skouras AZ, Kanellopoulos AK, Stasi S, Triantafyllou A, Koulouvaris P, Papagiannis G, Papathanasiou G. Clinical Significance of the Static and Dynamic Q-angle. Cureus. 2022 May 11;14(5):e24911. doi: 10.7759/cureus.24911. eCollection 2022 May. PMID 35698708
- [Derived] Lashien SA, Abdelnaeem AO, Gomaa EF. Effect of hip abductors training on pelvic drop and knee valgus in runners with medial tibial stress syndrome: a randomized controlled trial. J Orthop Surg Res. 2024 Oct 29;19(1):700. doi: 10.1186/s13018-024-05139-3. PMID 39468623